CLINICAL TRIAL: NCT07306442
Title: Abadan University of Medical Sciences
Brief Title: VR for Pain & Sleep in Burn Patients: A RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abadan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Rasool Paygozar, PhD student in Health Sciences, Faculty Member, Abadan University of Medical Sciences, Abadan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2004
Record Dates: First submitted 2025-12-04; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Burns; Pain; Sleep Disturbances
Keywords: Virtual reality; Non-pharmacological intervention; Wound dressing; Tbsa
MeSH Terms: conditions — Burns; Pain; Parasomnias | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group, randomized controlled trial comparing virtual reality intervention with standard care in burn patients.
Masking Description: Blinding was not feasible due to the visible nature of the VR headset and the need for participants and care providers to be aware of group assignment during the intervention. However, data collection and analysis were performed by blinded personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Intervention Group (Experimental): Participants in this group received immersive virtual reality distraction during their wound dressing change procedure. They wore an Oculus Quest 2 headset and were immersed in a calming, interactive virtual environment (e.g., a peaceful beach or forest) for the duration of the dressing change (approximately 30-45 minutes). The audio was enabled to enhance immersion.
  Interventions: Behavioral: Virtual Reality Distraction; Other: Standard Care
- Standard Care Group (Placebo Comparator): Participants in this group received standard care during their wound dressing change, which included verbal reassurance and routine analgesic administration as prescribed, without any additional distraction techniques such as virtual reality.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Virtual Reality Distraction — Participants in the experimental group received immersive virtual reality distraction during their wound dressing change procedure. They wore an Oculus Quest 2 headset and were immersed in a calming, interactive virtual environment (e.g., a peaceful beach or forest) for the duration of the dressing change (approximately 30-45 minutes). The audio was enabled to enhance immersion. This intervention aimed to reduce procedural pain and improve sleep quality through cognitive distraction and relaxation.
  Other Names: VR Therapy
  Arms: Virtual Reality Intervention Group
Other: Standard Care — Participants in the control group received standard care during their wound dressing change, which included verbal reassurance and routine analgesic administration as prescribed, without any additional distraction techniques such as virtual reality. No specific intervention was administered beyond standard clinical practice.
  Other Names: Routine Burn Care

SUMMARY:
This study aims to evaluate whether virtual reality (VR) can reduce pain and improve sleep quality during wound dressing changes in burn patients with 25-60% total body surface area (TBSA) burns, compared to standard care.

DETAILED DESCRIPTION:
Background:

Burn injuries are extremely painful, especially during wound dressing changes. They also cause severe sleep problems, which can slow down healing. While medicines help, they often have side effects and don't fully solve these issues. Virtual reality (VR) is a new tool that distracts the brain from pain by immersing patients in a calming digital world. This study was designed to assess if VR could help with both pain and sleep in burn patients.

Methods:

We conducted a randomized controlled trial with 60 adult burn patients who had between 25% and 60% of their body burned. All patients were stable and able to understand instructions. We randomly assigned them into two groups: one group used VR headsets during their dressing changes, and the other group received standard care without VR. Pain was measured before and after the procedure using a simple 0-to-10 scale. Sleep quality was assessed using a standard questionnaire (PSQI) before and 24 hours after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* - Adult patients aged 18 to 60 years.
* Deep partial-thickness or full-thickness burns covering 25% to 60% of total body surface area (TBSA).
* Hemodynamic stability (systolic BP ≥90 mmHg, HR 60-100 bpm, no vasopressor use).
* Ability to understand and comprehend Persian language.
* Scheduled for at least one standardized, non-sedated wound dressing change procedure.

Exclusion Criteria:

* - Diagnosed psychiatric or neurological disorder (e.g., schizophrenia, epilepsy).
* Severe visual impairment (best-corrected visual acuity <20/200) or auditory impairment.
* History of motion sickness or VR intolerance.
* Contraindications to VR use (e.g., active vertigo, uncontrolled hypertension).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) Total Score | 24 hours post-intervention
  The primary outcome for sleep quality was the change in the total score of the Pittsburgh Sleep Quality Index (PSQI) from baseline to 24 hours post-intervention. The PSQI is a validated self-report questionnaire assessing seven components of sleep quality over the past month. A higher score indicates poorer sleep quality. The change score (post-intervention minus pre-intervention) was calculated, with negative values indicating improvement.
Change in Visual Analog Scale (VAS) Pain Score | Immediately before and after the dressing change procedure
  The primary outcome for pain was the change in the Visual Analog Scale (VAS) score from immediately before to immediately after the wound dressing change procedure. The VAS is a 10-cm scale where 0 represents "no pain" and 10 represents "worst pain imaginable." The change score (post-procedure minus pre-procedure) was calculated, with negative values indicating pain reduction.

SECONDARY OUTCOMES:
Change in individual components of the Pittsburgh Sleep Quality Index (PSQI) | 24 hours post-intervention
  Secondary outcomes included changes in each of the seven individual components of the PSQI: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. These were assessed at baseline and 24 hours post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Taleghani Burn and Trauma Hospital, Ahvāz, Khuzestan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Yes, but only for specific purposes or under certain conditions Individual participant data (IPD) will be made available upon reasonable request to the corresponding author. Data sharing is subject to approval by the Ethics Committee of Abadan University of Medical Sciences and may require a formal data use agreement. Requests should include a detailed research proposal and must comply with local ethical and legal regulations.
Time Frame: Within 6 months after publication
Access Criteria: Request must include a detailed research proposal and be approved by the Ethics Committee of Abadan University of Medical Sciences

REFERENCES:
- [Background] Hoffman HG, Chambers GT, Meyer WJ 3rd, Arceneaux LL, Russell WJ, Seibel EJ, Richards TL, Sharar SR, Patterson DR. Virtual reality as an adjunctive non-pharmacologic analgesic for acute burn pain during medical procedures. Ann Behav Med. 2011 Apr;41(2):183-91. doi: 10.1007/s12160-010-9248-7. PMID 21264690
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771